CLINICAL TRIAL: NCT01979471
Title: The Alberta Vascular Risk Reduction Community Pharmacy Project: RxEACH
Acronym: RxEACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health & Wellness (Other Government); Alberta Health services (Other); Merck Frosst Canada Ltd. (Industry)
Responsible Party: Principal Investigator, Ross T. Tsuyuki, Professor of Medicine (Cardiology) and Director, EPICORE Centre University of Alberta, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: pro00041644
Record Dates: First submitted 2013-11-01; First posted 2013-11-08 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Diabetes; Chronic Kidney Disease; Established Atherosclerotic Vascular Disease; Framingham Risk Score More Than 20 Percent
Keywords: Cardiovascular risk reduction; Diabetes; Chronic Kidney Disease; Atherosclerotic vascular disease; Community Pharmacist; Randomized controlled trial; [eGFR <60 ml/min/1.73m2 and/or (ACR >= 30 mg/mmol or two consecutive ACR tests which are >= 3 mg/mmol)]
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Advanced care (Other): For all the patients randomized to the advanced care group the pharmacist will complete a Comprehensive Annual Care Plan (CACP) or Standard Medication Management Assessment (SMMA)
  Interventions: Other: Advanced Care
- Usual Care (No Intervention): Patients randomized to the usual care group will receive:
  * Usual pharmacy care with no specific interventions for 3 months
  * At the end of the 3 months of the usual care period, all patients will cross over to receive the advanced care outlined above for 3 months

INTERVENTIONS:
Other: Advanced Care — The pharmacist will complete a Comprehensive Annual Care Plan (CACP) or Standard Medication Management Assessment (SMMA), which will include:
  * Patient assessment
  * Laboratory assessment of HbA1c and lipids
  * Individual assessment of CVD risk and education about this risk
    * Calculation of cardiovascular risk will be facilitated by an online tool
    * Discussion of CVD risk with the patient using the interactive online tool which explains his/her individual cardiovascular risk and targets for intervention and providing the patient with education on cardiovascular risk factors and healthy lifestyle options
  * Treatment recommendations, Prescription adaptation(s), and/or prescribe where necessary to meet lipid, blood pressure and glycemic control targets and smoking cessation.
  * Regular communication with the patient's family physician after each contact with the patient
  * Regular follow-up with all patients a minimum of every 3-4 weeks for 3 months.
  Arms: Advanced care

SUMMARY:
Cardiovascular disease (disease of the heart and blood vessels) is one of the leading causes of death in Canada. It also carries a financial burden on the Canadian economy with a yearly cost close to $21 billion divided between loss of productivity and healthcare costs. The majority of cardiovascular disease cases (90%) are caused by factors that can be controlled and modified. These factors include high blood pressure, high cholesterol, diabetes (high blood sugar), tobacco smoking, unhealthy diet, obesity, physical inactivity and high alcohol consumption. Such factors are very common and not very well controlled and so individuals who have any of these factors would be at risk of having cardiovascular disease. As such controlling these factors will reduce the risk of having cardiovascular disease and improve the individuals' quality of life. Pharmacists frequently work with patients and their family doctor to provide cardiovascular care. Having a pharmacist involved in cardiovascular care may help patients with cardiovascular disease or at risk of having the disease because they are more accessible and may have more opportunities to educate people about cardiovascular medications. This might lead to better prevention and control of cardiovascular disease.

Purpose:

The research study will assess if a community pharmacy cardiovascular risk reduction intervention can help reduce cardiovascular risk.

Procedure:

If the individual has an elevated blood pressure, cholesterol, blood sugar, waist circumference or body weight or is physically inactive, have an unhealthy diet, a smoker or taking medications for any of the previously mentioned conditions, the pharmacist will assess the cardiovascular disease risk [risk of having a cardiovascular event (e.g. heart attack or a stroke)] using a computer program. If the individual is at high risk s/he will be asked to take part in the study.

If the individual agrees to take part in the study s/he will be randomly assigned to either the Usual Care Group or the Advanced Care Group. All participants have an equal chance of being assigned to either group. If assigned to the Usual Care Group, the individual will receive the care and services that would normally be provided by the pharmacist. At 3 months, the pharmacist will see the individual who will be offered the Advanced Care at that time.

If assigned to the to Advanced Care Group, the individual will be asked to meet with the pharmacist every 3-4 weeks over a 3 month period. During these meetings, the pharmacist will conduct an assessment that may include blood pressure, waist circumference, height and weight measurements and talk to the individual about their cardiovascular risk and medications. The individual and the pharmacist will come up with a plan for how to try to lower his/her cardiovascular risk. The pharmacist will discuss this plan with their family doctor. The individual will be asked to conduct some laboratory tests before the 3 months visit; these tests may include HbA1c (a blood test to measure blood sugar control over the last 3 months) and cholesterol to assess the effect of the intervention on cardiovascular risk.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death worldwide accounting for nearly one third of the total deaths. The majority (90%) of the CVD cases are caused by modifiable risk factors. These factors include tobacco smoking, hypertension, hyperlipidemia, diabetes, physical inactivity, high fat diet and obesity.

In Canada CVD rates have decreased drastically over the last few decades, yet it is still one of the leading causes of death. It also carries a financial burden on the Canadian economy with a cost close to $ 21 billion every year divided between loss of productivity and healthcare costs.

Despite the risks associated with the major CVD risk factors and the treatment advancement, their prevalence is still substantial in North America. Treatment gaps were also reported amongst such factors. Al Hamarneh and colleagues (2012) reported that almost 50% of the community dwelling patients with type 2 diabetes were not at their HbA1c target. Leiter and colleagues (2013) reported that almost half of the patients with type 2 diabetes did not achieve their HbA1c or cholesterol target, slightly more than one third achieved their blood pressure targets and only 13% achieved the composite triple target.

The guidelines recommend using cardiovascular risk assessment equations to guide CVD prevention and management. Despite being recommended by the guidelines, it has not been integrated in the clinicians' daily routine; in fact the majority of the patients attending physicians' clinics reported that they have never had a cardiovascular risk assessment. This indicates the need for new avenues for the patients to get their cardiovascular risk assessed.

Community pharmacists are front-line primary healthcare professionals who see patients with chronic diseases more frequently than family physicians; as such, they are well positioned to identify patients at high risk for CVD, determine their CVD risk and assist in their disease management. The efficacy of pharmacists' intervention in chronic disease has been well demonstrated in the literature. Two of the largest randomized controlled trials in community pharmacy setting were conducted by our group. Both studies reported positive impact of the pharmacist intervention on the patients' lipid panel and blood pressure.

Objectives

Primary objective

To evaluate the effect of a community pharmacy-based case finding and intervention program in patients at high risk for cardiovascular events on reduction in estimated risk for major cardiovascular events.

Secondary objectives

Clinical:

* Improvements in individual risk factors: LDL-cholesterol, blood pressure, HbA1c (among patients with diabetes), and smoking cessation
* Achievement of recommended cholesterol, blood pressure and glycemic control targets
* Increase in proportion of patients receiving appropriate BP, cholesterol and diabetes medication

Process:

* Increase in number of high risk patients screened for cardiovascular risk
* Assess the efficacy of various case-finding mechanisms and vulnerable patient population reach
* Assure sustainability by exploring enabling and barrier forces.

Methods

Design: Randomized controlled trial with patients as the unit of randomization

Setting: Community pharmacists in Alberta for recruitment and follow up, engaging both patients and family physicians

Patients/Population:

Inclusion criteria:

Adults (≥18 years of age) at high risk for cardiovascular events, including:

* Patients with diabetes
* Patients with chronic kidney disease [eGFR <60 ml/min/1.73m2 and/or (ACR >= 30 mg/mmol or two consecutive ACR tests which are >= 3 mg/mmol)]
* Patients with established atherosclerotic vascular disease including cerebrovascular disease (prior stroke or transient ischemic attack), cardiovascular disease (myocardial infarction, acute coronary syndrome, stable angina, or revascularization), or peripheral arterial disease (symptomatic and/or ankle brachial index <0.9).
* Primary prevention patients with multiple risk factors and Framingham risk score >20%
* In order to qualify for inclusion, all patients must have at least one uncontrolled risk factor (i.e., blood pressure, LDL-cholesterol, HbA1c, or current smokers.

Exclusion criteria:

* Unwilling to participate/sign consent form
* Unwilling or unable to participate in regular follow-up visits
* Pregnancy

Recruitment:

Pharmacists and pharmacy staff are going to use the following methods to recruit patients in the study:

· Proactive recruitment by case-finding facilitators (trained pharmacy technicians, assistants or pharmacy/medical/nursing students who focus on target prescriptions for oral hypoglycemic, anti-hypertensive and lipid lowering medications). Pharmacists will check the most recent lab results for those patients in the course of routine care. If the patient has not had an eGFR or proteinuria test done over the last 12 months he/she will be given a request to do those tests with a copy sent to his/her family physician.

If the Patient meets the inclusion criteria for the study the patient will be asked if he/she wants to participate in the study. If the patient agrees on participating he/she will be asked to sign a written informed consent form. After signing the consent form the patient will be enrolled in the study.

The patient's family physician is going to receive a letter from the pharmacist to inform him/her that his/her patient agreed to participate in this study.

Randomization:

Once informed written consent is obtained, the patients will be randomized (via a centralized secure website to ensure allocation concealment) in a 1:1 ratio to either advanced care or usual care groups

Intervention:

For all the patients randomized to the advanced care group the pharmacist will complete a Comprehensive Annual Care Plan (CACP) or Standard Medication Management Assessment (SMMA), which will include:

* Patient assessment (blood pressure measurement according to CHEP guidelines, waist circumference, weight and height measurements)
* Laboratory assessment of HbA1c and lipids (if not done within 3 months)
* Individual assessment of CVD risk and education about this risk

  * Calculation of cardiovascular risk will be facilitated by an online tool in which the pharmacist enters patient demographics such as age, gender, cholesterol, blood pressure, smoking status, diabetes, etc and the system will use the appropriate risk engine based on the patient's medical history. UKPDS, International model to predict recurrent cardiovascular disease and Framingham will be used for patients with diabetes, previous vascular disease, CKD or high Framingham risk (>20%) respectively (see appendix for risk engines score sheets). In the case where a patient has more than one co-morbidity the risk engine estimating the highest risk will be used
  * Discussion of CVD risk with the patient using the interactive online tool which explains his/her individual cardiovascular risk and targets for intervention
  * Proving the patient with education on cardiovascular risk factors and healthy lifestyle options
* Providing treatment recommendations (C-CHANGE and up to date Canadian clinical practice guidelines)
* Prescription adaptation(s), and/or prescribe where necessary to meet lipid, blood pressure and glycemic control targets and smoking cessation.
* Regular communication with the patient's family physician after each contact with the patient using the physician contact form which will be developed by the research team
* Regular follow-up with all patients a minimum of every 3-4 weeks for 3 months (Interim telephone follow-up may be performed at the discretion of the pharmacist; however telephone follow-up cannot be used for 2 consecutive visits or for the final visit (3 months).

Usual care:

Patients randomized to the usual care group will receive:

* Usual pharmacy care with no specific interventions for 3 months
* At the end of the 3 months of the usual care period, all patients will cross over to receive the advanced care outlined above for 3 months

The analysis of the results from patients who cross over from the usual care group into the advanced care group will be conducted separately on before and after design basis.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age) at high risk for cardiovascular events, including:

  * Patients with diabetes
  * Patients with chronic kidney disease [eGFR <60 ml/min/1.73m2 and/or (ACR >= 30 mg/mmol or two consecutive ACR tests which are >= 3 mg/mmol)]
  * Patients with established atherosclerotic vascular disease including cerebrovascular disease (prior stroke or transient ischemic attack), cardiovascular disease (myocardial infarction, acute coronary syndrome, stable angina, or revascularization), or peripheral arterial disease (symptomatic and/or ankle brachial index <0.9).
  * Primary prevention patients with multiple risk factors and Framingham risk score >20%
  * In order to qualify for inclusion, all patients must have at least one uncontrolled risk factor (i.e., blood pressure, LDL-cholesterol, HbA1c, or current smoking)

Exclusion Criteria:

* Unwilling to participate/sign consent form
* Unwilling or unable to participate in regular follow-up visits
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 723 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The difference in change in estimated cardiovascular risk between advanced care and usual care groups | 3 months
  The difference in change in estimated cardiovascular risk between advanced care and usual care groups

SECONDARY OUTCOMES:
Difference in change in individual cardiovascular risk factors between advanced care and usual care groups | 3 months
  Difference in change in individual cardiovascular risk factors between advanced care and usual care groups, including LDL-cholesterol, systolic and diastolic blood pressure, HbA1c, lifestyle (diet and exercise) and smoking cessation.
Achievement of individual and the "triple target" | 3 months
  Achievement of individual and the "triple target" of LDL-cholesterol ≤ 2.0 mmol/L, blood pressure control BP <140/90 mmHg (<130/80 in those with diabetes) and glycemic control (HbA1c ≤ 7.0) in advanced care compared to usual care group patients in those with diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte A Jones, MD, PhD, Principal Investigator — University of British Columbia - Southern Medical Program; Brenda Hemmelgarn, MD, PhD, Principal Investigator — Department of Medicine, University of Calgary; Ross T Tsuyuki, PharmD, MSc, Principal Investigator — Department of Medicine, University of Alberta
Locations (1):
- EPICORE Centre, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Tsuyuki RT, Al Hamarneh YN, Jones CA, Hemmelgarn BR. The Effectiveness of Pharmacist Interventions on Cardiovascular Risk: The Multicenter Randomized Controlled RxEACH Trial. J Am Coll Cardiol. 2016 Jun 21;67(24):2846-54. doi: 10.1016/j.jacc.2016.03.528. Epub 2016 Apr 4. PMID 27058907
- See also: Related Info — https://www.epicore.ualberta.ca/home/rxeach/